CLINICAL TRIAL: NCT06974149
Title: The Effects of Transcranial Direct Current Stimulation Associated With Neurofunctional Rehabilitation in Individuals With Spinocerebellar Ataxias - Randomized Clinical Trial
Brief Title: Effects of Transcranial Direct Current Stimulation Associated With Neurofunctional Rehabilitation in Individuals With Spinocerebellar Ataxias
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fernanda Cechetti, clinical professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUHSPortoAlegreMarianaBrutto
Record Dates: First submitted 2025-04-24; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Spinocerebellar Ataxia - All Sub-types
Keywords: spinocerebellar ataxias; transcranial direct current stimulation; neurological rehabilitation.
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- transcranial direct current stimulation associated with neurofunctional rehabilitation (Active Comparator)
  Interventions: Other: Neurofunctional Rehabilitation; Device: transcranial direct current stimulation
- transcranial direct current stimulation simulated associated with neurofunctional rehabilitation (Sham Comparator)
  Interventions: Other: Neurofunctional Rehabilitation; Device: transcranial direct current stimulation

INTERVENTIONS:
Other: Neurofunctional Rehabilitation — Neurofunctional Rehabilitation Protocol will consist of balance, motor coordination and gait exercises for 40 minutes and associated with tdcs
  Arms: transcranial direct current stimulation associated with neurofunctional rehabilitation
Device: transcranial direct current stimulation — Transcranial direct current stimulation will be applied for 20 minutes at an intensity of 2 mA. The anode will be placed on the scalp over the cerebellar area (2 cm below the inion); the cathode, in turn, will be placed on the spinal column in the lumbar enlargement (2 cm below T11)
  Arms: transcranial direct current stimulation associated with neurofunctional rehabilitation
Other: Neurofunctional Rehabilitation — Neurofunctional Rehabilitation Protocol will consist of balance, motor coordination and gait exercises for 40 minutes and associated with tdcs
  Arms: transcranial direct current stimulation simulated associated with neurofunctional rehabilitation
Device: transcranial direct current stimulation — Transcranial direct current stimulation will be applied for 30 seconds at an intensity of 2 mA. The anode will be placed on the scalp over the cerebellar area (2 cm below the inion); the cathode, in turn, will be placed on the spinal column in the lumbar enlargement (2 cm below T11). However the electrodes will be kept for 20 minutes to mask the stimulation
  Arms: transcranial direct current stimulation simulated associated with neurofunctional rehabilitation

SUMMARY:
The aim of this study is to evaluate the effects of . Transcranial direct current stimulation (tDCS) combined with neurofunctional rehabilitation on disease severity in individuals with neurodegenerative ataxias. The study will compare whether the Neurofunctional Rehabilitation Protocol combined with real tDCS will bring better results in reducing disease severity compared to the neurofunctional rehabilitation protocol combined with simulated tDCS.

DETAILED DESCRIPTION:
Neurodegenerative ataxias are a group of heterogeneous and progressive diseases that affect the cerebellum. Symptoms related to these diseases include difficulties with walking, balance, and motor coordination. Neurofunctional rehabilitation can help improve these motor symptoms. However, it is still limited in reducing neurodegeneration. Transcranial direct current stimulation (tDCS) applied to the cerebellum has shown to be a promising treatment in reducing disease severity, improving balance, and improving the quality of life of these individuals. tDCS in combination with neurofunctional rehabilitation may be a beneficial alternative in neurodegenerative ataxias, but studies are lacking. Regarding neurofunctional rehabilitation, some studies have shown improvements in reducing the progression of this pathology. However, as a rule, these studies presented poorly detailed protocols. Furthermore, the study populations included several types of cerebellar ataxias. Therefore, a detailed description of physiotherapy exercises, also recording them in images, with a more homogeneous sample, can ensure the viability of a more efficient treatment. tDCS applied to ataxia, in turn, presented beneficial results regarding disease progression, walking speed, balance and, also, quality of life. tDCS can enhance the effects of neurofunctional rehabilitation, as has already been proven in other populations. The combination of tDCS with neurofunctional rehabilitation is still poorly described in the literature in patients with neurodegenerative ataxias. Therefore, it is necessary to conduct a study specifically designed to test the hypothesis that tDCS combined with neurofunctional rehabilitation will demonstrate better results in relation to disease severity, postural control, risk of falls, quality of life and fatigue. In this case, a ten-session protocol can be applied, evaluating the results in 5 (five) ,10 (ten) and 20 (twenty)sessions, positioning the anode in the cerebellum and the cathode in the spinal cord, with patient monitoring for 16 (sixteen) weeks. This study can, finally, compare the results between neurofunctional rehabilitation combined with tDCS and neurofunctional rehabilitation alone

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spinocerebellar ataxias;
* Walking independently or with aids;

Exclusion Criteria:

* Metal implants in the brain or spinal column and Cochlear implants;
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) | baseline, at the end of 5 ,10 and 20 sessions and follow up ( 2 and 4 months)
  The severity of ataxia will be assessed using the Ataxia Rating and Assessment (SARA) scale, which consists of eight items: gait, posture, sitting, speech, finger-chasing, nose-finger test, rapid alternation of hand movements, and lower limb coordination. The higher the score, the greater the severity of the disease.

SECONDARY OUTCOMES:
Mini-BEST test | baseline, at the end of 5 ,10 and 20 sessions and follow up ( 2 and 4 months)
  The Mini-BEST is an instrument that assesses postural control. The Mini-BEST includes 14 items divided into: anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. The following tasks will be assessed: sitting to standing, standing on tiptoe, single-leg support, correction with anterior, posterior, and lateral steps, eyes open on a firm surface, eyes closed on an unstable surface, tilt with eyes closed, change in gait speed, walking with head turns, walking and turning on the axis, passing through obstacles, gait speed with and without dual task. The individual may use an assistive device during the test, if necessary, but each domain will be scored one level below the item for which the device was used . The maximum score is 28 (twenty-eight) points; Items can be scored as 0 (unable),
Stabilometry | baseline, at the end of 5 ,10 and 20 sessions and follow up ( 2 and 4 months)
  Stabilometry assesses balance in the orthostatic posture and quantifies the anteroposterior and lateral oscillations of the body's center of pressure (COP). This analysis will be performed using a Baiobit inertial sensor (BTS Bioengineering). The sensor will be connected to the individual by an elastic belt placed at the height of the S1-S2 vertebrae. The patient will remain in a bipedal position for 30 (thirty) seconds. The sensor will measure the following indices: angle of oscillations, elliptical area, oscillations, speed of anteroposterior and lateral oscillations of the center of mass and the length of the trajectory of the center of mass.
Falls Efficacy Scale-International (FES-I) | baseline, at the end of 5,10 and 20 sessions and follow up ( 2 and 4 months)
  This scale assesses the risk of falls. It is a questionnaire of self-efficacy and confidence in balance, with 16 (sixteen) items. It includes questions about activities of daily living in the home environment and in the community environment. Response options include: not at all concerned, somewhat concerned, very concerned and extremely concerned.
  The score ranges from a minimum of 16 (no concern about falls) to a maximum of 64 (severe concern about falls). Therefore, the higher the score, the greater the risk of falls.
Timed Up and Go (TUG) | baseline, at the end of 5 ,10 and 20 sessions and follow up ( 2 and 4 months)
  The Timed Up Go (TUG) test will be used to assess functional mobility and the risk of falls. The test identifies the speed at which the patient can get up from a chair, walk 3 (three) meters, return and sit down. The time spent performing the task can be classified as low risk, medium risk and high risk of falls. During the test, the patient will be wearing a Baiobit inertial sensor (BTS Bioengineering). The sensor will be connected to the individual by an elastic belt placed at the height of the S1-S2 vertebrae. This sensor will assess the duration of the TUG phases (sitting to standing, walking, turning and standing to sitting).
8-meter walk test (8mWT) | baseline, at the end of 5,10 and 20 sessions and follow up ( 2 and 4 months)
  The 8-meter walk test is a functional assessment that measures an individual's walking speed. The test will be performed indoors on a flat surface, on a path marked out at 8 meters. Adhesive tape will be used to clearly mark the start and end of the path, and a stopwatch will be used to measure walking time. Individuals will be instructed to walk "as quickly but safely as possible." If necessary, individuals may use any assistive device, but without the help of another person or a wall. Three (3) repetitions will be performed, with a 1 (one) minute recovery interval between each repetition. The average time will be calculated and from this average the speed will be determined using the equation: Speed = distance traveled/time.
Gait analysis | baseline, at the end of 5,10 and 20 sessions e follow up ( 2 and 4 months)
  This analysis will be performed using a Baiobit inertial sensor (BTS Bioengineering). The sensor will be connected to the individual by an elastic belt placed at the height of the S1-S2 vertebrae. The individuals will be instructed to walk a distance of 7 meters. The following variables will be collected: speed (m/s), cadence (steps/min), stride length (meters), number of steps, stance phase (% of cycle) and swing phase (% of cycle).
Form Health Survey 36 (SF-36) | baseline, at the end of 5,10 and 20 sessions and follow up ( 2 and 4 months)
  Quality of life will be assessed using the Form Health Survey 36 (SF-36), a questionnaire consisting of 36 scores that assess 8 subdomains: vitality, limitation due to physical aspect, functional capacity, bodily pain, general health perceptions, social aspects, emotional aspects and mental health . This instrument has been translated and culturally validated for the Brazilian population . It presents a score from 0 to 100, in which zero corresponds to the "worst general health status" and 100 the "best general health status" .
Modified Fatigue Impact Scale (MFIS) | baseline, at the end of 5 ,10 and 20 sessions and follow up ( 2 and 4 months)
  The Modified Fatigue Impact Scale (MFIS) is a scale that assesses fatigue. It consists of 21 statements that assess the physical, cognitive and psychosocial domains. The individual must choose an alternative (scored from 0 to 4) for each item. Possible answers include: "never", "rarely", "rarely", "often" and "always". To answer it, the last two weeks up to the present day must be considered. The total MFIS score ranges from 0 to 84 and is calculated by adding the statements. Its objective is to assess the impact of fatigue on the patient's life. Values below 38 correspond to the absence of fatigue. For scores equal to or greater than 38, the higher the score, the greater the impact of fatigue